CLINICAL TRIAL: NCT06200701
Title: Intervention Program of a Job Crafting: Job Crafting Behavior, Work Meaningfulness, Change Attitude, Task and Adaptive Performance Among Nurses
Brief Title: Intervention Program of a Job Crafting
Acronym: JobCrafting
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: IRB0001123
Record Dates: First submitted 2023-12-26; First posted 2024-01-11 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2023-12

CONDITIONS: Educational Problems; Work-Related Condition; Nurse's Role

STUDY DESIGN:
Who Masked: Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Program application of a Job Crafting (Experimental): job crafting training program designed for this study was implemented through twelve sessions, from which three theory and nine practical sessions were held in a room at the worksite. The sessions were conducted outside of working hours in the hospital These sessions lasted 21 hours; 3 theory hours (one hour for each theoretical session); and 9 practical sessions (two hours for each practical session). Having the whole number of nurses at the same time was difficult, so the nurses were classified into five groups each group consisting of about 16 nurses. All sessions were repeated to the five main groups until 80 nurses completed the entire 21-hours instruction period
  Interventions: Behavioral: Job Crafting program
- non Intervention Program application (No Intervention): non Intervention Program application

INTERVENTIONS:
Behavioral: Job Crafting program — The training program designed for this study was implemented through twelve sessions, from which three theory and nine practical sessions were held in a room at the worksite. The sessions were conducted outside of working hours in the hospital These sessions lasted 21 hours; 3 theory hours (one hour for each theoretical session); and 9 practical sessions (two hours for each practical session). Having the whole number of nurses at the same time was difficult, so the nurses were classified into five groups each group consisting of about 16 nurses. All sessions were repeated to the five main groups until 80 nurses completed the entire 21-hours instruction period
  Arms: Intervention Program application of a Job Crafting

SUMMARY:
The implementation of effective intervention programs is crucial in enhancing the overall well-being and performance of healthcare professionals, particularly in demanding environments such as nursing

DETAILED DESCRIPTION:
The implementation of effective intervention programs is crucial in enhancing the overall well-being and performance of healthcare professionals, particularly in demanding environments such as nursing. This study focuses on the design and impact of an intervention program centered around job crafting among nurses. Job crafting involves employees proactively shaping their roles to align with personal strengths and preferences. In the context of nursing, this intervention aims to investigate the influence of job crafting behavior on various dimensions, including work meaningfulness, change attitude, task performance, and adaptive performance. Understanding the interplay between job crafting and these critical aspects is essential for developing targeted strategies to improve job satisfaction, performance, and adaptability among nurses, ultimately contributing to the enhancement of overall healthcare quality. This introduction sets the stage for exploring the multifaceted effects of a job crafting intervention within the nursing profession.

ELIGIBILITY:
Inclusion Criteria:

* willingness to participate
* less than 60 years old

Exclusion Criteria:

* enter training in any educational program at least 6 months

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 160 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-01-30 (Estimated)

PRIMARY OUTCOMES:
nurses' job crafting | three months
  Nurses who were exposed to the job crafting program exhibited a higher score in job crafting by job crafting questionnaire (total score of job crafting questionnaire ( 13-65) and higher score in Job Crafting questionnaire (26-65) than nurses who were not exposed
nurses' Work And Meaning | three months
  nurses who were exposed to the job crafting program exhibited a higher score in Work Meaning attitude by Work And Meaning Inventory (total score range from 10-50 and higher score from 20 to 50)

CONTACTS AND LOCATIONS:
Overall Officials: mohamed H atta, Study Director — Faculty of nursing, Alexandria university, Egypt
Locations (1):
- Faculty of Nursing, Masjid al Khiḑr, Semoha, Egypt

DOCUMENTS (1):
  • Study Protocol (2024-01-08): https://cdn.clinicaltrials.gov/large-docs/01/NCT06200701/Prot_000.pdf